CLINICAL TRIAL: NCT03691636
Title: A Single Center, Randomized, Controlled Trial Evaluating the Efficacy and Safety of Eyelash Prostheses Compared to 5.0% Lifitegrast Ophthalmic Solution in Subjects With Dry Eye Disease.
Brief Title: Eyelash Prostheses Compared to 5.0% Lifitegrast BID for Dry Eye Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: D.E.L., LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D.E.L. 002
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Eyelash Prostheses (Experimental): Each subject in this arm will receive eyelash prostheses according to a specified algorithm by a certified eyelash extensions.
  Interventions: Device: Eyelash prostheses
- 5.0% Lifitegrast Ophthalmic Solution (Active Comparator): Each subject in this arm will receive 5.0% Lifitegrast eye drops BID
  Interventions: Device: 5.0% Lifitegrast Ophthalmic Solution

INTERVENTIONS:
Device: Eyelash prostheses — Eyelash prostheses are essentially specialized eyelash extensions
  Arms: Eyelash Prostheses
Device: 5.0% Lifitegrast Ophthalmic Solution — 5.0% Lifitegrast Ophthalmic Solution
  Arms: 5.0% Lifitegrast Ophthalmic Solution

SUMMARY:
This is a single-center, randomized, controlled trial to evaluate the safety and efficacy of eyelash prostheses versus 5.0% Lifitegrast BID, in 40 patients (20 randomized to each of two arms of the study) evaluated at 3 weeks and 5 weeks, respectively, after initiation of treatment.

DETAILED DESCRIPTION:
This is a single center, randomized, controlled clinical trial to evaluate the tolerability, efficacy, and safety of eyelash prostheses over a 3-week period versus Xiidra BID over a 5 week period in subjects with self-reported DED. 40 subjects will be randomized to either eyelash prostheses or Xiidra, in a 1:1 ratio.

At Visit 1 (screening), informed consent will be obtained from subjects and eligibility will then be determined. All pre-treatment assessments will be done at this visit. Randomization will occur. If randomized to receive Xiidra eye drops, a prescription will be written and the treatment will be started right away. If randomized to eyelash prostheses, then a second study visit will be made approximately 2 weeks later.

Visit 2 (Eyelash Prostheses application) Subjects randomized to receive eyelash prostheses will have them applied approximately 2 weeks after the screening and randomization visit.

Visit 3 (Final visit) will be 3 weeks post eyelash prosthesis placement and 5 weeks post Xiidra eye drop initiation. This was done to compare the maximal treatment effect between the two groups. All subjects will undergo post-treatment assessments.

At each visit, patients will be asked to report any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported dry eye symptoms
2. Tear Break Up Time of less than 10 seconds as assessed by the Oculus Keratograph (see Appendix A).
3. SPEED II Score greater than 25
4. Men or Women, age between 50 and 90 inclusive
5. Willingness to undergo both pre-treatment and post-treatment testing per the protocol
6. Willingness to endure the 2-3 hour time required to place eyelash extensions, if randomized to this treatment arm
7. Willingness to use eye drops for dry eyes and fill a prescription through insurance coverage, if randomized to this treatment arm
8. Willingness to attend all study visits
9. Willingness to sign informed consent and liability waiver

   -

Exclusion Criteria:

1. Absence of eyelashes
2. Eyelash disease such as clinically significiant demodex, blepharitis, meibomitis
3. Be unable or unwilling to give written informed consent and/or to comply with study procedures.
4. Have any known hypersensitivity or contraindication to study treatments (including excipients), topical anesthetics or vital dyes.
5. Be unable to demonstrate correct instillation of over the counter (OTC) ocular lubricant during Visit 1.
6. Have clinically significant ocular surface disease in either eye (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with study safety procedures, or assessments.
7. Have clinically significant systemic disease (e.g., uncontrolled diabetes, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study at Visit 1 and 2.
8. Current use of Restasis or Xiidra at the time of Visit 1
9. Changes in the dose of, or the initiation of, any medications that are known to affect dry eyes within 90 days of Visit 1 or during the duration of the study.
10. Any history of Herpes simplex of Herpes zoster affecting the eye or head.

    -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-02 (Estimated); Primary Completion 2019-04-02 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferior change from baseline in tear break up time as measured by the Oculus Keratograph in the interventional subjects compared to the active control subjects | The primary endpoint will be assessed 3 weeks after eyelash prosthesis placement in the interventional arm and 5 weeks after initiation of eye drops in the active comparator arm
  A non-inferiority endpoint in tear break up time

SECONDARY OUTCOMES:
Non-inferior change in tear meniscus height as measured by the Oculus Keratograph in the treatment subjects compared to control subjects | The secondary endpoint will be assessed 3 weeks after eyelash prosthesis placement in the interventional arm and the interventional arm and 5 weeks after initiation of eye drops in the active comparator arm
  Non-inferiority endpoint in tear meniscus height
Non-inferior change from baseline in SPEED II questionnaire in the treatment subjects compared to the control subjects | The secondary endpoint will be assessed 3 weeks after eyelash prosthesis placement in the interventional arm and the interventional arm and 5 weeks after initiation of eye drops in the active comparator arm
  Non-inferiority endpoint in the SPEED II questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Korenfeld, MD, Principal Investigator — Comprehensive Eye Care
Locations (1):
- Comprehensive Eye Care, Washington, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data